CLINICAL TRIAL: NCT01035034
Title: Comparison of "One-stop" Hybrid Coronary Revascularization Versus Percutaneous Coronary Intervention for the Treatment of Multi-vessel Coronary Artery Disease
Brief Title: Comparison of One-stop Hybrid Revascularization Versus Percutaneous Coronary Intervention for the Treatment of Multi-vessel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: China National Center for Cardiovascular Diseases ( Shengshou Hu MD, FACC ), China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20091217
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2009-12-21 (Estimated); Status verified 2009-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- One-stop hybrid coronary revasularization (Experimental): Percutaneous Coronary Intervention; Coronary Artery Bypass
  Interventions: Procedure: Hybrid MIDCAB/PCI
- PCI with stenting (Active Comparator): Percutaneous Coronary Intervention
  Interventions: Procedure: PCI with DES

INTERVENTIONS:
Procedure: Hybrid MIDCAB/PCI — MIDCAB with no associated or concomitant surgical procedures, using partial ministernotomy, without cardiopulmonary bypass (CPB) and cardioplegia. PCI with drug eluting stents (DES) performed by cardiologists on the non-LAD lesions in the same operating suite immediately following MIDCAB.
  Device: Polymer-based Sirolimus-Eluting Stents (SES).
  Arms: One-stop hybrid coronary revasularization
Procedure: PCI with DES — Polymer-based Sirolimus-Eluting Stents (SES)
  Arms: PCI with stenting

SUMMARY:
The "one-stop" hybrid coronary revascularization combines minimally invasive direct coronary artery bypass (MIDCAB) and PCI to be performed in the hybrid operating suite, an enhanced operating room equipped with radiographic capability. This study is to compare 1-year clinical outcomes of "one-stop" hybrid coronary revascularization with percutaneous coronary intervention (PCI) in selected patients with multivessel coronary artery disease.

DETAILED DESCRIPTION:
Rationale and purpose of this study:

"One-stop" (also named simultaneous) hybrid coronary revascularization has emerged as a novel, safe and feasible minimally invasive approach in selected patients with multivessel coronary artery disease (CAD). The benefits of "one-stop" hybrid procedure compared with conventional PCI are unclear, however.

This study is a single center randomized clinical trial to compare the safety and efficacy of "one-stop" hybrid procedure with conventional PCI in the treatment of selected patients with multivessel CAD requiring revascularization with suitable coronary anatomy.

Sample size:

We examined the results of SYNTAX trial and of the hybrid procedures published previously. The 1-year MACCE rate (the primary endpoint) is estimated as being 18% for PCI/stenting and 8% for the hybrid group. The sample calculated for this trial is 480 patients.

Design/Methodology:

Trial design: A single center randomized clinical trial comparing "one-stop" hybrid procedure versus conventional PCI with SES in 480 patients with suitable anatomy who need revascularization.

Intervention: Patients will be randomized to undergo either "one-stop" hybrid procedure or conventional PCI with SES.

Randomization:

Patients will be evaluated by both a cardiac surgeon and an interventional cardiologist. After obtaining informed written consent, patients will be randomized to receive "one-stop" hybrid procedure or conventional PCI with SES. An expertise-based randomization will be used.

The data adjudicators will be blinded to the study. Due to the nature of this study, the operating surgeons, cardiologists, anesthetists, other operative room staff, and ICU staff will not be blind in this study.

Study intervention:

Candidates will be randomized to receive "one-stop" hybrid procedure or conventional PCI.

ELIGIBILITY:
Inclusion Criteria:

* Two- or three-vessel disease, left main disease, or LM equivalent with 2 or 3-vessel disease (left anterior descending [LAD], left circumflex [LCX], right coronary artery [RCA] territory)
* Denovo lesions of LAD , with obstruction >=70%, especially chronic totally occlusion (CTO), severe calcification or bifurcation lesion of the LM;
* Angiographic characteristics of non-LAD lesion(s) amiable to PCI/stenting;
* Chronic stable or unstable angina pectoris of CCS 2 or greater (symptoms of angina and/or objective evidence of myocardial ischemia);
* Evaluated by both cardiac surgeon and cardiologist together.

Exclusion Criteria:

* Need for emergent CABG;
* Prior CABG;
* Prior PCI with stenting within 6 months of study entry;
* Stroke with 6 months of study entry;
* Overt congestive heart failure;
* Need for a concomitant operation (i.e. valve repair or replacement, Maze surgery);
* Hemodynamic instability;
* Situations in which complete revascularization is not possible served;
* Allergy to radiographic contrast, aspirin or clopidogrel.
* Contradictions to PCI: Occluded coronary vessels, PVD, Unable to achieve access, Fresh thrombus, Vessels <1.5mm; Intolerance to aspirin or both clopidogrel and ticlopidine;
* Cannot undergo either CABG or PCI/DES because of a coexisting medical condition
* History of significant bleeding; Significant leukopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2009-12; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Composite of major adverse cardiac or cerebrovascular events (MACCE) including death, myocardial infarction, stroke and/or repeat revascularization. | 1 year

SECONDARY OUTCOMES:
Overall MACCE rate. | 30 days after procedure and 2 years after enrollment
Cardiac death. | 30 days after procedure, 1 and 2 years after enrollment
Documented myocardial infarction. | 30 days after procedure, 1 and 2 years after enrollment
Target lesion revascularization. | 30 days after procedure, 1 and 2 years after enrollment
Recurrence of Angina. | 1 and 2 years after enrollment
Cost-effectiveness analysis. | 1 and 2 years after enrollment
Quality of life. | 6 months, 1 and 2 years after enrollment
Rehospitalization. | 6 months, 1 and 2 years after enrollment
Stent thrombosis. | 30 days after procedure, 6 months, 1 and 2 years after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Shengshou Hu, M.D., Study Director — China National Center for Cardiovascular Diseases
Locations (2):
- China (2):
  - China National Center for Cardiovascular Diseases, Cardiovascular Institute & Fuwai Hospital, Beijing, Beijing Municipality
  - Institute of cardiovascular diseases & Fuwai hospital, Beijing, Beijing Municipality